CLINICAL TRIAL: NCT00872898
Title: An Open-label (Part One) and a Randomized, Double-blind, Placebo-Controlled (Part Two) Study of the Pharmacokinetics, Safety, Efficacy, and Tolerability of Memantine in Pediatric Patients With Autism
Brief Title: Study of Pharmacokinetics, Safety, Efficacy, and Tolerability of Memantine in Children With Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEM-MD-57A
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-11

CONDITIONS: Autism
Keywords: autism; memantine; pediatric; Forest Laboratories; Autism in pediatric patients
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Once daily oral administration of memantine for 12 weeks.
  Interventions: Drug: Memantine - Extended Release (ER)
- 2 (Placebo Comparator): Once daily oral administration of placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine - Extended Release (ER) — Memantine - 3mg and 6mg capsules, dose ranging 3 - 18 mg/day in 4 weight groups, administered orally.
  Other Names: Namenda ER
  Arms: 1
Drug: Placebo — Placebo capsules, once daily, oral administration.
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of memantine extended release, as well as its extent of absorption in pediatric patients with autism.

DETAILED DESCRIPTION:
This is a multicenter, two-part study in pediatric (ages 6 to 18 years) patients diagnosed with autism.

Patients participating in Part One will receive a single open-label dose of memantine. Blood samples for pharmacokinetic analysis will be collected.

Part Two is a randomized, double-blind, placebo-controlled 12-week efficacy and safety study evaluating change in all core domains (social interactions, communication, and restricted interests and repetitive behaviors) of autism.

In the Forest autism trials conducted in children ages 6-12, dosing with an extended release formulation of memantine was weight-based. These weight based dose limits were selected to ensure exposure in terms of area under the curve (AUC) was less than the predefined limit of 2100 ng∙h/mL that represented a 10-fold lower exposure than observed at the NOAEL (No observed adverse effect level) of 15 mg/kg/day in juvenile rats.

The weight-based dose limits in these studies were as follows:

* Group A: ≥ 60 kg; max 15 mg/day
* Group B: 40-59 kg; max 9 mg/day
* Group C: 20-39 kg; max 6 mg/day
* Group D: < 20 kg; max 3 mg/day

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 6 to 12 years
* Diagnosis of autistic disorder, according to DSM-IV-TR using Autism Diagnostic Interview-Revised and Autism Diagnostic Observation Schedule (modules 2 & 3).
* A knowledgeable caregiver capable of providing reliable information about the patient's condition, able to attend all clinic visits with the patient
* Patients over age 12, only if they completed Study MEM-PK-21

Exclusion Criteria:

* Medical history of active epilepsy/seizure disorder except simple febrile seizures
* Participation in any other clinical investigation using an experimental drug within 30 days of the start of this study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2009-04; Primary Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ephraim Katz, PhD, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories, Inc.
Locations (17):
- United States (17):
  - Forest Investigative Site, Phoenix, Arizona
  - Forest Investigative Site, Sacramento, California
  - Forest Investigative Site, San Francisco, California
  - Forest Investigative Site, Santa Ana, California
  - Forest Investigative Site, Stanford, California
  - Forest Investigative Site, Jacksonville Beach, Florida
  - Forest Investigative Site, St. Petersburg, Florida
  - Forest Investigative Site, Hoffman Estates, Illinois
  - Forest Investigative site, Naperville, Illinois
  - Forest Investigative Site, Indianapolis, Indiana
  - Forest Investigative Site, Cambridge, Massachusetts
  - Forest Investigative Site, Toms River, New Jersey
  - Forest Investigative Site, Voorhees Township, New Jersey
  - Forest Investigative Site, Manhasset, New York
  - Forest Investigative Site, Cleveland, Ohio
  - Forest Investigative Site, Columbus, Ohio
  - Forest Investigative Site, Oklahoma City, Oklahoma

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Brignell A, Marraffa C, Williams K, May T. Memantine for autism spectrum disorder. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013845. doi: 10.1002/14651858.CD013845.pub2. PMID 36006807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients for Part One of the study were recruited during a 15 month period from April of 2009, to June of 2010. Patients for Part Two of the study were recruited for a 37 month period from April of 2009 to April of 2012. All study sites were located in the United States.
Pre-assignment Details: Part One of the study enrolled 4 patients to determine a safe dosing regimen for Part Two. One patient from Part One of the study also enrolled in Part Two. The 121 patients enrolled in Part Two were randomized after two weeks of single-blind placebo treatment.
Groups:
- Placebo: Once daily, oral administration of placebo for 12 weeks.
- Memantine: Once daily oral administration of memantine extended release for 12 weeks.
  Memantine - 3mg and 6mg capsules, dose ranging 3 - 18 mg/day in 4 weight groups, administered orally.
Period: Part One - Open Label, Pharmacokinetics
Arm/Group | Placebo | Memantine
Started | 0 | 4
Completed | 0 | 4
Not Completed | 0 | 0
Period: Part Two - Double Blind
Arm/Group | Placebo | Memantine
Started | 61 | 60
Completed | 50 | 54
Not Completed | 11 | 6
Not completed — Adverse Event | 4 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Other reasons | 2 | 0

BASELINE CHARACTERISTICS:
Population: Part One of the study enrolled 4 patients to determine a safe dosing regimen for Part Two along with data collected for 14 patients enrolled in study MEM-PK-21. One patient from Part One of the study also enrolled in Part Two. The 121 patients enrolled in Part Two were randomized after two weeks of single-blind placebo treatment.
Groups:
- Part One - Memantine: Patients received a single dose of 3-mg memantine extended release capsule, oral administration.
- Part Two - Placebo: Once daily oral administration of placebo for 12 weeks.
- Part Two - Memantine: Once daily oral administration of memantine extended release for 12 weeks. Memantine - 3mg and 6mg capsules, dose ranging 3 - 18 mg/day in 4 weight groups.
- Total: Total of all reporting groups
Arm/Group | Part One - Memantine | Part Two - Placebo | Part Two - Memantine | Total
Number analyzed (Participants) | 3 | 61 | 60 | 124
Age, Continuous [Mean (Standard Deviation); unit: years]
  6 years to 18 years | 9.0 (2.6) | 8.9 (2.2) | 9.0 (2.2) | 9.0 (0.1)
Age, Customized [Number; unit: participants]
  6 years to 12 years | 3 | 60 | 59 | 122
  13 years to 18 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 12 | 8 | 22
  Male | 1 | 49 | 52 | 102
Region of Enrollment [Number; unit: participants]
  United States | 3 | 61 | 60 | 124

OUTCOME MEASURES:

1. Primary Outcome: Extent of Absorption of Memantine (Part One)
Description: Area under the plasma concentration vs. time curve (AUC) for memantine, as measured in units of nanogram x hours per milliliter.
Time Frame: Baseline to 144 hours. Measurements were taken 0 (predose), 4, 8, 24, 30, 48, 96 and 144 hours post-dose
Population: Four patients enrolled in Part One, receiving a single dose of memantine and having evaluable pharmacokinetic parameters (Pharmacokinetic Population)
Measure: Mean (Standard Deviation); unit: ng•h/mL
Groups:
- Memantine: Patients received a single dose of 3-mg memantine extended release capsule, oral administration.
Arm/Group | Memantine
Number analyzed (Participants) | 4
ng•h/mL | 682.53 (217.77)

2. Secondary Outcome: Core Autism Treatment Scale-Improvement: Total Score
Description: The Core Autism Treatment Scale-Improvement (CATS-I) is based on rating 14 items from 1 (very much improved) to 7 (very much worse) with a total score ranging from 14 (improved) to 98 (worsened).
  The Core Autism Treatment Scale-Improvement (CATS-I) is designed to utilize a comparison between pretreatment ratings of Core Autism Treatment Scale-Severity (CATS-S) and ratings of improvement after start of therapy (CATS-I). Both parts of the CATS contain 14 items testing for social interaction (items 1-9) and communication (items 10-14). Each of these items is rated from 1 (indicating most benign) to 7 (indicating most severe).
Time Frame: At Week 12
Population: All of the the 121 randomized patients in Part Two of the study, received at least 1 dose of study drug. The protocol specified Intent-to-Treat (ITT) Population consisted of 107 patients who had at least 1 postbaseline assessment of SRS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Once daily oral administration of placebo for 12 weeks.
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | 50.4 (1.0) | 48.3 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.1197, mixed-model for repeated measures; Least squares mean difference = -2.2, 95% CI 2-sided [-4.9 to 0.6]

3. Primary Outcome: Change in Total Raw Score of Social Responsiveness Scale
Description: The Social Responsiveness Scale (SRS) is a 65-item informant-rated assessment, ranging from 0 (no impairment) to 195 (severe social impairment).
  Each item is associated with 1 of 5 subscales (social awareness, social cognition, social communication, social motivation and autistic mannerisms). Each item is rated on a 4-point scale from 1 (not true) to 4 (almost always true). The scores are then transposed to a scale from 0 to 3 and scores are summed within each of the 5 subscales. A higher score indicates greater severity of social impairment.
Time Frame: From Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | -9.5 (2.6) | -9.6 (2.5)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.9781, mixed-model for repeated measures; Least squares mean difference = -0.1, 95% CI 2-sided [-7.2 to 7.0]

4. Secondary Outcome: Core Autism Treatment Scale-Improvement: Social Interaction
Description: The Core Autism Treatment Scale-Improvement (CATS-I) Social Interaction Subscale is based on rating 9 items from 1 (very much improved) to 7 (very much worse) with a total score ranging from 9 (improved) to 63 (worsened).
  The Core Autism Treatment Scale-Improvement (CATS-I) is designed to utilize a comparison between pretreatment ratings of Core Autism Treatment Scale-Severity (CATS-S) and ratings of improvement after start of therapy (CATS-I). Both parts of the CATS contain 14 items testing for social interaction (items 1-9) and communication (items 10-14). Each of these items is rated from 1 (indicating most benign) to 7 (indicating most severe).
Time Frame: At Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | 32.4 (0.7) | 31.1 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.1459, mixed-model for repeated measures; Least squares mean difference = -1.4, 95% CI 2-sided [-3.2 to 0.5]

5. Secondary Outcome: Core Autism Treatment Scale-Improvement: Communication
Description: The Core Autism Treatment Scale-Improvement (CATS-I) Communication Subscale is based on rating 5 items from 1 (very much improved) to 7 (very much worse) with a total score ranging from 5 (improved) to 35 (worsened).
  The Core Autism Treatment Scale-Improvement (CATS-I) is designed to utilize a comparison between pretreatment ratings of Core Autism Treatment Scale-Severity (CATS-S) and ratings of improvement after start of therapy (CATS-I). Both parts of the CATS contain 14 items testing for social interaction (items 1-9) and communication (items 10-14). Each of these items is rated from 1 (indicating most benign) to 7 (indicating most severe).
Time Frame: At Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | 18.0 (0.4) | 17.2 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.1344, mixed-model for repeated measures; Least squares mean difference = -0.8, 95% CI 2-sided [-1.9 to 0.3]

6. Secondary Outcome: Change in Children's Communication Checklist-2 (CCC-2) - Speech Subscale
Description: The Children's Communication Checklist-2 (CCC-2) Speech Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
  The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties children may have (across 10 different subscales, consisting of 7 items each) that affect communication (items 1-50), as well as strengths that children may demonstrate when communicating with others (items 51-70).
Time Frame: From Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | -0.4 (0.5) | -0.7 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.7000, mixed-model for repeated measures; Least squares mean difference = -0.2, 95% CI 2-sided [-1.5 to 1.0]

7. Secondary Outcome: Change in Children's Communication Checklist-2 (CCC-2) - Syntax Subscale
Description: The Children's Communication Checklist-2 (CCC-2) Syntax Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
  The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties children may have (across 10 different subscales, consisting of 7 items each) that affect communication (items 1-50), as well as strengths that children may demonstrate when communicating with others (items 51-70).
Time Frame: From Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | -1.1 (0.4) | -1.2 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.9069, mixed-model for repeated measures; Least squares mean difference = -0.1, 95% CI 2-sided [-1.3 to 1.1]

8. Secondary Outcome: Change in Children's Communication Checklist-2 (CCC-2) - Semantics Subscale
Description: The Children's Communication Checklist-2 (CCC-2) Semantics Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
  The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties children may have (across 10 different subscales, consisting of 7 items each) that affect communication (items 1-50), as well as strengths that children may demonstrate when communicating with others (items 51-70).
Time Frame: From Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | -0.2 (0.3) | -0.5 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.4679, mixed-model for repeated measures; Least squares mean difference = -0.3, 95% CI 2-sided [-1.2 to 0.6]

9. Secondary Outcome: Change in Children's Communication Checklist-2 (CCC-2) - Coherence Subscale
Description: The Children's Communication Checklist-2 (CCC-2) Coherence Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
  The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties children may have (across 10 different subscales, consisting of 7 items each) that affect communication (items 1-50), as well as strengths that children may demonstrate when communicating with others (items 51-70).
Time Frame: From Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | -1.2 (0.5) | -1.2 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.9598, mixed-model for repeated measures; Least squares mean difference = -0.0, 95% CI 2-sided [-1.3 to 1.3]

10. Secondary Outcome: Change in Children's Communication Checklist-2 (CCC-2) - Initiation Subscale
Description: The Children's Communication Checklist-2 (CCC-2) Initiation Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
  The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties children may have (across 10 different subscales, consisting of 7 items each) that affect communication (items 1-50), as well as strengths that children may demonstrate when communicating with others (items 51-70).
Time Frame: From Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | -0.8 (0.5) | -0.9 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.9898, mixed-model for repeated measures; Least squares mean difference = -0.0, 95% CI 2-sided [-1.3 to 1.3]

11. Secondary Outcome: Change in Children's Communication Checklist-2 (CCC-2) - Scripted Language Subscale
Description: The Children's Communication Checklist-2 (CCC-2) Scripted Language Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
  The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties children may have (across 10 different subscales, consisting of 7 items each) that affect communication (items 1-50), as well as strengths that children may demonstrate when communicating with others (items 51-70).
Time Frame: From Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | -1.0 (0.4) | -0.5 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.4228, mixed-model for repeated measures; Least squares mean difference = 0.5, 95% CI 2-sided [-0.7 to 1.6]

12. Secondary Outcome: Change in Children's Communication Checklist-2 (CCC-2) - Context Subscale
Description: The Children's Communication Checklist-2 (CCC-2) Context Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
  The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties children may have (across 10 different subscales, consisting of 7 items each) that affect communication (items 1-50), as well as strengths that children may demonstrate when communicating with others (items 51-70).
Time Frame: From Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | -1.5 (0.4) | -0.2 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.0201, mixed-model for repeated measures; Least squares mean difference = 1.4, 95% CI 2-sided [0.2 to 2.5]

13. Secondary Outcome: Change in Children's Communication Checklist-2 (CCC-2) - Nonverbal Communication Subscale
Description: The Children's Communication Checklist-2 (CCC-2) Nonverbal Communication Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
  The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties children may have (across 10 different subscales, consisting of 7 items each) that affect communication (items 1-50), as well as strengths that children may demonstrate when communicating with others (items 51-70).
Time Frame: From Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | -0.7 (0.4) | -0.9 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.6889, mixed-model for repeated measures; Least squares mean difference = -0.2, 95% CI 2-sided [-1.3 to 0.9]

14. Secondary Outcome: Change in Children's Communication Checklist-2 (CCC-2) - Social Relations Subscale
Description: The Children's Communication Checklist-2 (CCC-2) Social Relations Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
  The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties children may have (across 10 different subscales, consisting of 7 items each) that affect communication (items 1-50), as well as strengths that children may demonstrate when communicating with others (items 51-70).
Time Frame: From Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | -1.0 (0.4) | -0.8 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.7481, mixed-model for repeated measures; Least squares mean difference = 0.2, 95% CI 2-sided [-0.9 to 1.2]

15. Secondary Outcome: Change in Children's Communication Checklist-2 (CCC-2) - Interests Subscale
Description: The Children's Communication Checklist-2 (CCC-2) Interests Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
  The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties children may have (across 10 different subscales, consisting of 7 items each) that affect communication (items 1-50), as well as strengths that children may demonstrate when communicating with others (items 51-70).
Time Frame: From Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 53 | 54
units on a scale | -0.5 (0.4) | -0.5 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Memantine; Test type: Superiority or Other; p = 0.9500, mixed-model for repeated measures; Least squares mean difference = -0.0, 95% CI 2-sided [-1.2 to 1.1]

ADVERSE EVENTS:
Time Frame: Adverse event data for Part One of this study was collected over a 14-month period from May 2009 to July of 2010. Adverse event data for Part Two of this study was collected over a 38-month period from July of 2009 to September of 2012.
Groups:
- Placebo - Part Two, Double-Blind Treatment: Once daily oral administration of placebo for 12 weeks
- Memantine - Part Two, Double-Blind Treatment: Once daily oral administration of memantine extended release for 12 weeks.
  Memantine - 3mg and 6mg capsules, dose ranging 3 - 18 mg/day in 4 weight groups.
- Memantine - Part One, Open Label Treatment: Patients received a single dose of 3-mg memantine extended release capsule, oral administration.
Arm/Group | Placebo - Part Two, Double-Blind Treatment | Memantine - Part Two, Double-Blind Treatment | Memantine - Part One, Open Label Treatment
Serious Adverse Events (participants affected / at risk) | 0/61 | 1/60 | 0/4
Other Adverse Events (participants affected / at risk) | 31/61 | 37/60 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Part Two, Double-Blind Treatment (N=61) | Memantine - Part Two, Double-Blind Treatment (N=60) | Memantine - Part One, Open Label Treatment (N=4)
Affective Disorder (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Part Two, Double-Blind Treatment (N=61) | Memantine - Part Two, Double-Blind Treatment (N=60) | Memantine - Part One, Open Label Treatment (N=4)
Headache (Nervous system disorders) | 3 | 3 | 1
Vomiting (Gastrointestinal disorders) | 6 | 4 | 0
Irritability (General disorders) | 3 | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 6 | 0
Influenza (Infections and infestations) | 2 | 4 | 0
Psychomotor hyperactivity (Nervous system disorders) | 4 | 1 | 0
Aggression (Psychiatric disorders) | 3 | 5 | 0
Agitation (Psychiatric disorders) | 1 | 4 | 0
Insomnia (Psychiatric disorders) | 3 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0
Anxiety (Nervous system disorders) | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 2 | 0
Pyrexia (General disorders) | 4 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study are the property of Forest Research Institute. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute.